CLINICAL TRIAL: NCT00204867
Title: CT Virtual Colonoscopy for Primary Colorectal Screening
Brief Title: Virtual Colonoscopy (VC) for Primary Colorectal Screening
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Naval Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 2004-0104
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Polyps
Keywords: colorectal; polyps
MeSH Terms: conditions — Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: In vivo surveillance of 6-9 mm polyps detected at CTC
  Interventions: Other: CTC surveillance

INTERVENTIONS:
Other: CTC surveillance — In vivo CTC surveillance of 6-9 mm polyp

SUMMARY:
This study involves a primary VC screening for colorectal polyps. The research hypothesis is that VC screening, including surveillance of sub-cm polyps, is a safe and effective approach.

DETAILED DESCRIPTION:
The purpose of this study is to use virtual colonoscopy screening to learn more about what happens to small colon polyps (less than 10 mm) over time. From this, we can find out whether it's safer to remove all colon polyps right away or leave the small ones in place and remove only those that grow to 10 mm or more.

ELIGIBILITY:
Inclusion Criteria:

* Medium-sized colorectal polyps (6-9 mm)

Exclusion Criteria:

* No medium-sized colorectal polyps (6-9 mm)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Screening population for colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2004-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The growth rate (natural history) of small colorectal polyps | The outcome measure of polyp growth rate is established at the time of surveillance CTC by comparing to the baseline CTC
  Polyp growth rates are established by comparing polyp volume at the initial and surveillance CTC studies

CONTACTS AND LOCATIONS:
Overall Officials: Perry J. Pickhardt, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Pickhardt PJ, Kim DH, Pooler BD, Hinshaw JL, Barlow D, Jensen D, Reichelderfer M, Cash BD. Assessment of volumetric growth rates of small colorectal polyps with CT colonography: a longitudinal study of natural history. Lancet Oncol. 2013 Jul;14(8):711-20. doi: 10.1016/S1470-2045(13)70216-X. Epub 2013 Jun 7. PMID 23746988